CLINICAL TRIAL: NCT05373498
Title: Pediatric Resuscitation Outcome in Children With Heart Disease
Brief Title: Resuscitation Registry in CHD
Acronym: PRO-CHD
Status: Recruiting | Type: Observational
Sponsor: Leipzig Heart Science gGmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other); Zentrum für Klinische Studien Leipzig (Other); Deutsche Gesellschaft für Pädiatrische Kardiologie und Angeborene Herzfehler e.V. (Unknown); Stiftung KinderHerz (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-0450
Record Dates: First submitted 2022-03-25; First posted 2022-05-13 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest; Congenital Heart Disease
Keywords: pediatric resuscitation outcome; congenital heart disease; neurodevelopmental outcome
MeSH Terms: conditions — Heart Arrest; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children with congenital heart defects are far more likely to suffer a cardiovascular arrest and be in the need of cardiopulmonary resuscitation than healthy children or those with diseases of other organ systems, especially after cardiothoracic surgery. Due to a lack of data, the exact number of resuscitations in this patient cohort, as well as the morbidity and mortality, is unknown. This study aims to register all cardiovascular arrests in pediatric patients with congenital heart disease and study the mortality and morbidity with a special focus on the neurodevelopmental outcome.

DETAILED DESCRIPTION:
Background and aim: Children with heart defects, especially those after heart surgery, have an up to ten times higher risk for an in-hospital cardiac arrest, compared to children without heart disease. Although this patient cohort is particularly vulnerable, these events and outcomes are not systematically monitored in Germany. We designed a prospective multicenter-registry study aiming to record in-hospital cardiac arrests of children with congenital- (CHD) and acquired heart disease in Germany.

Methods: A web-based registry was designed, prospectively collecting data (patient´s demographics, CPR data, post-resuscitation care and clinical course, neurological outcome and follow-up), according to the Utstein template. All children (0-18 years) with heart disease suffering a cardiac arrest requiring resuscitation of ≥ two minutes will be included. The primary outcome is survival to discharge, the secondary outcome is morbidity, with a particular focus on neurological morbidity. An inclusion of 10-20 children/centre/year is anticipated. As this is an observational study, no intervention is planned.

Results: This registry will provide data on the mortality, early and mid-term neurologic outcome, and quality of life after cardiac arrest of children with heart disease in Germany. Correlations between patients´ characteristics, resuscitation characteristics and post-resuscitation care with primary and secondary outcomes will be analyzed.

Conclusions: By systematically recording and analyzing the outcome after in-hospital cardiac arrest in children with CHD, this study is an important first step to close knowledge gaps regarding the risk factors and outcome of cardiac arrest in this patient group, and aims to improve care and outcomes of these vulnerable patients.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart defects, congenital heart arrhythmia, familial cardiomyopathies, inflammatory heart diseases
* pediatric resuscitation (chest compressions ≥2min) in hospital or on arrival in hospital
* age <18 years
* informed consent of the parents or legal representative

Exclusion Criteria:

* absence or withdrawal of informed consent of the parents or legal representative
* do-not-resuscitate-order (DNR)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children: 0 - 18 years
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
survival to hospital discharge | until the date of discharge or death from any cause, whichever came first, assessed up to 2 months

SECONDARY OUTCOMES:
Number of return of spontaneous circulation | until the date of discharge or spontaneous circulation from any cause, whichever came first, assessed up to 2 months
Rate of morbidity | until 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Bonn (AöR), Bonn

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Markel F, Kramer P, Anand J, Heimberg E, Herbsleb V, Amann V, Herberg U, von Borell du Vernay F, Seidemann K, Liem L, Michaelis A, Schmitt K, Weidenbach M. Paediatric Resuscitation Outcome in Children with Heart Disease (ProCHD): protocol of a Germany-wide multicentre, prospective open registry. BMJ Open. 2026 Jan 8;16(1):e107163. doi: 10.1136/bmjopen-2025-107163. PMID 41506771